CLINICAL TRIAL: NCT00633542
Title: Thalidomide-Dexamethasone vs Alpha-Interferon-Dexamethasone as Maintenance Therapy After Thalidomide, Dexamethasone and Pegylated Liposomal Doxorubicin Combination for
Brief Title: Maintenance Therapy After Thalidomide-Dexamethasone(ThaDD) for Multiple Myeloma(MM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Offidani Massimo, Clinica di Ematologia Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO 02/02 MM; AIL 2002
Record Dates: First submitted 2008-01-02; First posted 2008-03-12 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Multiple Myeloma
Keywords: thalidomide; maintenance; interferon; dexamethasone; newly diagnosed multiple myeloma; relapsed refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD (Experimental): thalidomide-dexamethasone
  Interventions: Drug: thalidomide
- ID (Active Comparator): Interferon-dexamethasone
  Interventions: Drug: interferon alpha

INTERVENTIONS:
Drug: thalidomide — 100 mg/day orally until progression or severe toxicity
  Arms: TD
Drug: interferon alpha — 3 MU 3 times a week until progression or severe toxicity
  Arms: ID

SUMMARY:
This is randomized, multicentre study aimed to compare a standard maintenance therapy with Interferon-Dexamethasone with an experimental therapy based on Thalidomide-Dexamethasone in patients with multiple myeloma who responded to ThaDD induction therapy

DETAILED DESCRIPTION:
Thalidomide has already been used as maintenance and/or consolidation after high-dose therapy followed by autologous stem cell transplantation. Despite a number of phase II and III studies the issues of right dose and duration of thalidomide and subsets of patients benefiting from it have not yet been settled We explored the maintenance therapy after thalidomide, dexamethasone and pegylated liposomal doxorubicin called ThaDD protocol. Patients with de novo or relapsed MM obtaining at least minor response after 4 to 6 ThaDD courses, were randomized to receive standard maintenance therapy with IFN 3 MU 3 times a week or an experimental maintenance therapy such as thalidomide 100 mg per day until relapse or intolerable side effects. Both groups also received pulsed dexamethasone 20 mg 4 days a month.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed or advanced multiple myeloma achieving at least a minimal response after induction with ThaDD regimen
* Written consent

Exclusion Criteria:

* peripheral neuropathy >= grade 2
* neutropenia < 1000/mcl or thrombocytopenia < 50000/mcl
* severe depression
* organ disfunction > grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
progression free survival | 3 years

SECONDARY OUTCOMES:
overall survival safety | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Offidani Massimo, MD, Principal Investigator — clinica di ematologia ospedali riuniti ancona università politecnica delle marche; Pietro Leoni, MD, PhD, Study Chair — clinica di ematologia università politecnica delle marche
Locations (1):
- Clinica di ematologia ospedali riuniti ancona università politecnica delle marche, Ancona, Italy

REFERENCES:
- [Background] Offidani M, Corvatta L, Piersantelli MN, Visani G, Alesiani F, Brunori M, Galieni P, Catarini M, Burattini M, Centurioni R, Ferranti M, Rupoli S, Scortechini AR, Giuliodori L, Candela M, Capelli D, Montanari M, Olivieri A, Poloni A, Polloni C, Marconi M, Leoni P. Thalidomide, dexamethasone, and pegylated liposomal doxorubicin (ThaDD) for patients older than 65 years with newly diagnosed multiple myeloma. Blood. 2006 Oct 1;108(7):2159-64. doi: 10.1182/blood-2006-03-013086. Epub 2006 Jun 8. PMID 16763209